CLINICAL TRIAL: NCT07377136
Title: Studie Vlivu Urolithinu A na Populaci s BI vyšším neý 30 při výživové Restrikci
Brief Title: Influence of the Urolithin A on the Population With BMI Higher Than 30 During Restricted Eating.
Acronym: Obesity UroA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Pavel Borsky, Principal Investigator, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202509 P05
Record Dates: First submitted 2025-09-29; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Obesity & Overweight
Keywords: obesity; urolithinA; restricted eating
MeSH Terms: conditions — Obesity; Overweight | interventions — 3,8-dihydroxy-6H-dibenzo(b,d)pyran-6-one

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, randomized, placebo-controlled, parallel-group trial in adults aged 30-60 years with BMI >30 kg/m² and elevated visceral adiposity. Participants are randomized 1:1 to Urolithin A 500 mg once daily vs matching placebo for 24 weeks, on top of a standardized lifestyle program (individualized energy restriction with higher protein, reduced carbohydrates, time-restricted eating 11:13, and sleep-hygiene optimization). Randomization is stratified by sex (male/female) and age (≤45/≥45). Study visits include baseline, ~3-weekly follow-ups, and an end-of-study visit. Primary domain is preservation of functional muscle mass during weight loss; key secondary domains include body composition, cardiometabolic/inflammatory markers, mitochondrial/aging biomarkers, autonomic/vascular indices, and patient-reported outcomes.
Who Masked: Participant, Care Provider, Investigator
Masking Description: only those above
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Urolithin A (Experimental)
  Interventions: Dietary Supplement: Urolithin A 500mg

INTERVENTIONS:
Dietary Supplement: Urolithin A 500mg — Dietary Supplement: Urolithin A (500 mg) - Intervention Description Oral Urolithin A 500 mg capsule once daily for 24 weeks, preferably with the first meal. GMP-manufactured product; identical capsule shell/appearance to placebo. No dose titration. No other dietary supplements allowed during participation. Adherence assessed by pill counts and visit logs; temporary interruption permitted for adverse events per protocol. Co-administered with the same standardized lifestyle program as the control arm.
  Arms: Urolithin A
Other: Placebo — Placebo Comparator: Matching Placebo - Intervention Description Matching inert capsule (no Urolithin A), same size, color, shell, and packaging as active product; once daily for 24 weeks with the first meal. Dispensed in coded kits to maintain masking. Participants receive the same lifestyle program as the active arm. Use of other dietary supplements is prohibited during the trial.
  Arms: Placebo

SUMMARY:
Purpose. This study will test whether daily Urolithin A (500 mg) for 6 months helps adults with obesity lose weight while preserving functional muscle mass and improving markers of mitochondrial health, inflammation, and metabolism. All participants receive the same structured lifestyle program (nutrition and sleep guidance); half will receive Urolithin A and half a matching placebo.

Background. Weight loss can improve health but may also reduce skeletal muscle, especially in people with obesity. Aging and obesity are both linked to mitochondrial dysfunction, impaired autophagy/mitophagy, oxidative stress, and low-grade inflammation. Urolithin A is a gut-derived, diet-related compound that promotes mitophagy and may support muscle function and metabolic health.

Design. Single-center, randomized, placebo-controlled, parallel-group trial. About 100 adults aged 30-60 years with BMI >30 kg/m² and elevated visceral adiposity will be enrolled and randomized in a 1:1 ratio (stratified by sex and age ≤45 vs ≥45 years). Blinding will include participants, study staff, and assessors.

Intervention.

Urolithin A 500 mg orally once daily vs matching placebo, for 24 weeks.

A standardized lifestyle program for all participants: individualized energy restriction with higher protein intake, reduced carbohydrates, and time-restricted eating (11-hour eating window / 13-hour overnight fast); plus structured sleep-hygiene recommendations and light daily activity guidance.

No other dietary supplements are allowed during the study.

Main assessments. At baseline and regularly during the study, participants will undergo:

Body composition by bioimpedance (InBody), including skeletal muscle and visceral fat indices.

Muscle function (handgrip dynamometry; 30-second chair-stand).

Cardiometabolic and inflammatory biomarkers from blood (standard biochemistry, lipids, glucose/HbA1c, CRP; exploratory cytokines/adipokines).

Mitochondrial/aging biomarkers, including DNA-based epigenetic aging measures.

Cardiovascular/ANS function (heart-rate variability and vascular indices; MaxPulse Medicore).

Questionnaires on sleep quality, physical activity, and weight-management self-efficacy.

Visits and duration. 6-month participation with baseline, 3-weekly check-ins, and a final visit for repeat testing and blood sampling.

Outcomes. The study focuses on safety and on whether Urolithin A, compared with placebo, helps preserve functional muscle mass and improves mitochondrial, inflammatory, and metabolic biomarkers during weight loss.

Who can join. Adults 30-60 years with obesity and higher visceral fat who are willing to follow the lifestyle program. Key medical exclusions (e.g., diabetes, active autoimmune disease, pregnancy) and supplement restrictions apply; full criteria are provided in the Eligibility section.

Potential benefits and risks. Participants may benefit from weight loss support and close monitoring. Risks include blood draw discomfort and potential, usually mild, supplement-related side effects. Safety will be monitored throughout.

Location and sponsor. The study is conducted at Charles University, Faculty of Medicine in Hradec Králové (Czech Republic) under the Department of Preventive Medicine.

DETAILED DESCRIPTION:
Scientific Background and Rationale

Obesity and aging share pathophysiological features-mitochondrial dysfunction, impaired autophagy/mitophagy, oxidative stress, and chronic low-grade inflammation-that contribute to loss of skeletal muscle and functional capacity ("sarcopenic obesity") and increased frailty risk. While weight reduction improves cardiometabolic health, it can also decrease lean mass if not carefully managed.

Urolithin A (UA) is a bioactive metabolite derived from ellagitannins that has shown the ability to activate mitophagy, support mitochondrial function, and favor muscle health in preclinical and early clinical studies. We hypothesize that, when combined with a standardized lifestyle program, UA 500 mg/day will preserve functional muscle mass and favorable biomarker profiles during intentional weight loss in adults with obesity.

Objectives

Primary objective:

Evaluate the safety and efficacy of 6 months of Urolithin A 500 mg once daily versus placebo, in addition to a structured lifestyle program, in adults with obesity undergoing dietary restriction. Efficacy focuses on preservation of functional muscle mass in the context of weight loss and on improvements in biomarkers of mitochondrial function, inflammation, and metabolic health.

Key secondary objectives:

Quantify changes in body composition (skeletal muscle mass; visceral adiposity) over time.

Assess muscle strength and endurance (handgrip dynamometry; 30-second chair-stand).

Evaluate systemic inflammatory and oxidative-stress markers and metabolic profile (e.g., lipids, glucose/HbA1c, CRP).

Explore the impact on biological aging using validated epigenetic aging and related molecular biomarkers.

Characterize changes in autonomic/vascular indices (e.g., HRV, arterial elasticity) and patient-reported outcomes (sleep, activity, weight-management self-efficacy).

Examine associations between lifestyle adherence and outcomes.

Study Design

Prospective, single-center, randomized, placebo-controlled, parallel-group clinical trial with blinded participants, investigators, and outcome assessors. Target enrollment: ~100 participants (approximately balanced by sex and age group ≤45 vs ≥45 years via stratified randomization).

Arms and Interventions

Experimental (Urolithin A): Urolithin A 500 mg oral capsule once daily for 24 weeks.

Control (Placebo): Matching placebo capsule once daily for 24 weeks.

Co-intervention (both arms): A standardized lifestyle program tailored to baseline anthropometrics, comprising:

Energy restriction with higher protein intake (approx. 1.0-1.5 g/kg/day) and reduced carbohydrates; emphasis on minimally processed foods.

Time-restricted eating: 11-hour eating window with 13-hour overnight fast (e.g., ~08:00-19:00).

Sleep-hygiene optimization: regular bed/wake times; targets of 7.5-9 hours of nightly sleep; guidance on environment, light exposure, stimulants, and pre-sleep routines.

Light daily activity guidance. Use of other dietary supplements is prohibited during participation.

Schedule of Assessments

Screening / "Visit 0": Eligibility review; bioimpedance to confirm visceral fat level threshold; anthropometry; blood pressure.

Baseline (Day 0): Informed consent; questionnaires; blood sampling; bioimpedance (InBody); MaxPulse Medicore autonomic/vascular testing; muscle strength (handgrip dynamometry, average of 3 trials + peak value) and muscle endurance (30-second chair-stand); individualized nutrition and sleep-hygiene education.

Follow-ups: Approximately every 3 weeks-anthropometry, blood pressure, bioimpedance, MaxPulse Medicore, muscle testing, adherence review, and lifestyle adjustments as needed.

End of Study (Week 24): Repeat baseline assessments and final blood sampling; exit interview.

Outcome Domains (entered in detail in the Outcomes module)

Functional muscle preservation: bioimpedance-derived skeletal muscle indices; handgrip strength; chair-stand repetitions.

Body composition: total fat mass; visceral adipose area/score; segmental lean/fat distribution.

Cardiometabolic/Inflammatory biomarkers: standard biochemistry (electrolytes, liver/kidney function, lipids, glucose/HbA1c, CRP) and exploratory panels (e.g., TNF-α, IL-6, adipokines, myostatin, SIRT1, endothelial adhesion molecules).

Mitochondrial/healthy aging measures: DNA-based epigenetic aging clocks and related molecular markers from whole blood.

Autonomic/vascular function: HRV metrics, arterial elasticity, and vascular flow indices via MaxPulse Medicore.

Patient-reported outcomes: sleep quality (PSQI), physical activity (GPAQ), and weight-management self-efficacy (WEL).

Eligibility (summary; see Eligibility module for full criteria)

Adults 30-60 years with BMI >30 kg/m² and elevated visceral fat by bioimpedance who can follow the lifestyle program. Key exclusions include thyroid disease, type 2 diabetes, autoimmune/inflammatory bowel disease, active malignancy, pregnancy/lactation or planned pregnancy, severe psychiatric disease limiting adherence, major uncontrolled comorbidities, significant musculoskeletal limitations, and use of dietary supplements other than the study product.

Randomization, Blinding, and Allocation Concealment

Participants will be randomized 1:1 to UA or placebo using a computer-generated sequence with stratification by sex and age. Identical capsules will be dispensed to maintain blinding of participants, site staff, and assessors. Emergency unblinding procedures will be in place.

Safety Monitoring

Adverse events (AEs), vitals, and laboratory parameters will be collected at each visit. Women of child-bearing potential will follow pregnancy precautions; pregnancy during the study leads to discontinuation of the investigational product and withdrawal from the trial. Pre-specified stopping rules include serious or unexpected adverse reactions deemed related to the study product. AEs/SAEs will be recorded and reported per applicable regulations.

Concomitant Medications and Prohibited Therapies

Stable chronic medications are permitted when clinically necessary; major changes (e.g., for hypertension) are allowed only as needed and will be documented. All non-study dietary supplements are prohibited during participation.

Adherence and Retention

Adherence will be supported through structured education, 3-weekly check-ins, and review of pill counts and lifestyle logs (nutrition, sleep, activity). Motivational elements include a brief written statement of goals at baseline.

Biospecimen Handling

Blood samples will be pseudonymized and processed according to standard operating procedures for clinical chemistry/hematology, ELISA panels (inflammation, adipokines, etc.), and DNA extraction for epigenetic analyses. Samples will be delivered to designated laboratories within defined processing windows.

Statistical Considerations

Analyses will follow intention-to-treat with a per-protocol sensitivity set. Continuous outcomes will be analyzed using ANCOVA or mixed-effects models with baseline values and stratification factors as covariates. Categorical outcomes will use appropriate models (e.g., χ² or logistic regression). Pre-specified subgroup analyses by sex and age group will be performed. With ~100 participants, the study is powered to detect a moderate effect size in body-composition/functional endpoints while characterizing safety and biomarker trajectories.

Ethics and Oversight

The protocol will receive Ethics Committee/IRB approval prior to enrollment. The trial will be conducted in accordance with the Declaration of Helsinki and Good Clinical Practice. All participants will provide written informed consent. Data confidentiality will be maintained using coded identifiers and secure storage.

Expected Impact

If effective, Urolithin A could provide a simple, adjunctive strategy to protect muscle health and improve biological aging and metabolic markers during dietary weight loss in adults with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-60 years (inclusive) at screening
* BMI > 30 kg/m² at screening
* Visceral fat level ≥ 12 by segmental bioimpedance (InBody) at screening
* Able and willing to follow the standardized lifestyle program (individualized energy restriction with higher protein, reduced carbohydrates, time-restricted eating 11:13) and sleep-hygiene guidance for 24 weeks
* Willing to attend baseline and ~3-weekly follow-ups; undergo blood draws, bioimpedance, MaxPulse testing, and muscle strength/endurance tests; and complete questionnaires (WEL, PSQI, GPAQ)
* Medication stability: chronic medications (e.g., treated hypertension, antidepressants) stable for ≥3 months before baseline; only clinically necessary changes allowed during the study
* Permitted conditions/therapies (if stable): common allergies/atopic eczema; food intolerances; contraception and menopausal hormone therapy
* Women of childbearing potential: negative pregnancy test at baseline; agreement to use highly effective contraception during the study and for 4 weeks after last dose; not breastfeeding
* Able to provide written informed consent

Exclusion Criteria:

* Known thyroid disease (untreated/unstable hypothyroidism or hyperthyroidism)
* Type 2 diabetes mellitus (diagnosed or on glucose-lowering therapy)
* Autoimmune disease, including psoriasis
* Inflammatory bowel disease or other chronic inflammatory GI disorders (e.g., Crohn's disease, celiac disease)
* Dyslipidemia treated with statins
* Pregnancy, lactation, or planned pregnancy during the study period
* Active malignant disease
* Cognitive impairment or neurodegenerative disease that may affect consent or adherence
* Severe psychiatric disorder that would preclude participation (e.g., severe major depression) or unstable depression/medication changes within the past 3 months
* Uncontrolled comorbidity or decompensated chronic disease (e.g., uncontrolled hypertension; systolic ≥175 mmHg at screening)
* Severe or limiting musculoskeletal condition preventing participation in assessments or the lifestyle program
* Use of non-study dietary supplements (vitamins, herbal/nutraceutical products) that the participant is unwilling or unable to discontinue from baseline through end of study
* Known allergy/intolerance to Urolithin A or capsule excipients
* Any condition that, in the investigator's judgment, makes participation unsafe or could compromise data integrity

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Appendicular Skeletal Muscle Index (ASMI) by Bioimpedance | Baseline to Week 24 (end of intervention)
  ASMI = sum of lean mass in both arms and legs (kg) divided by height² (m²), derived from segmental bioimpedance (InBody). Primary comparison is change from baseline to Week 24 between Urolithin A and placebo using ANCOVA adjusting for baseline, sex, and age stratum. Higher ASMI reflects greater functional muscle mass.

SECONDARY OUTCOMES:
Change in Handgrip Strength (kg) | Baseline to Week 24
  Dominant-hand grip strength measured with a calibrated handheld dynamometer; average of 3 trials (peak also recorded). Between-group difference in change from baseline to Week 24.
Change in Visceral Adipose Area (cm²) by Bioimpedance | Baseline to Week 24
  Visceral fat area (VFA, cm²) from InBody bioimpedance. Lower values indicate improvement. Between-group difference in change from baseline to Week 24.
Change in Percent Body Fat (%) | Baseline to Week 24
  Whole-body fat percentage by bioimpedance (InBody). Between-group difference in change from baseline to Week 24.
Glycemic Control (HbA1c) | Baseline to Week 24
  Change from baseline in HbA1c (%). Between-group difference (Urolithin A vs placebo) in change to Week 24 (ANCOVA with baseline, sex, age stratum).
LDL-C | Baseline to Week 24
  Change from baseline in LDL-C. Between-group difference in change to Week 24.
Inflammation (suPAR) | Baseline to Week 24
  Change from baseline in systemic inflammatory marker (suPAR; ng/mL). Between-group difference in change to Week 24.
GDF15 | Baseline to Week 24
  Change from baseline in serum GDF15 (assay units). Between-group difference in change to Week 24.
Autonomic/Vascular Function (Arterial Elasticity) | Baseline to Week 24
  Change from baseline arterial elasticity score (MaxPulse Medicore). Between-group difference in change to Week 24.
Epigenetic Aging Panel (DNA Methylation Age Acceleration) | Baseline to Week 24
  Change from baseline in blood-based DNA methylation age acceleration (years; difference between DNAm age and chronological age; pre-specified clocks). Between-group difference in change to Week 24.
Weight-Loss Responder Rates (≥5% and ≥10% Body Weight) | Baseline to Week 24
  Proportion of participants achieving ≥5% and ≥10% reduction from baseline body weight. Between-group comparison at Week 24.
Patient-Reported Outcomes Panel (WEL) | Baseline to Week 24
  Change from baseline in Weight Efficacy Lifestyle Questionnaire total score (WEL). Between-group difference in change to Week 24.
Patient-Reported Outcomes Panel (PSQI) | Baseline to Week 24
  Change from baseline in Pittsburgh Sleep Quality Index total score (PSQI). Between-group difference in change to Week 24.
Patient-Reported Outcomes Panel (GPAQ) | Baseline to week 24
  Change from baseline in Global Physical Activity Questionnaire total MET-minutes/week (GPAQ). Between-group difference in change to Week 24.
Safety Panel (TEAEs and SAEs) | From first dose to Week 24
  Participants with treatment-emergent adverse events and serious adverse events, coded by SOC/PT; severity and relatedness summarized by arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Charles University, Faculty of Medicine in Hradec Kralove, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: No